CLINICAL TRIAL: NCT00338429
Title: Better Days, Better Nights: Treatment for Sleep Difficulties (A Sleep Intervention Module of the Family Help Program)
Brief Title: Better Days, Better Nights: Treatment for Sleep Difficulties (Telephone Coached)
Acronym: Sleep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3104; NSHRF grant (Other: nshrf)
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Sleep Disorder
Keywords: sleep onset latency; bedtime resistance
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment: FHP Sleep Program (Experimental): Stratified with or without behavior Disorder Diagnosis (ADHD): 50% randomized to receive Better Days, Better Nights- sleep distance intervention
  Interventions: Behavioral: FHP Sleep Program
- Control: Usual Care (No Intervention): Stratified with/without behavior diagnosis (ADHD): 50% randomized to receive usual care for sleep disorder

INTERVENTIONS:
Behavioral: FHP Sleep Program — Cognitive-Behavioral Intervention
  Arms: Treatment: FHP Sleep Program

SUMMARY:
The purpose of the Strongest Families (formerly Family Help Program)is to evaluate the effectiveness of the Strongest Families distance intervention compared to usual or standard care that is typically provided to children with mild to moderate sleep onset latency and/or bedtime resistance difficulties. This is a single-centre trial based at the IWK Health Centre. The primary outcome is change in sleep patterns (sleep onset latency and/or bedtime resistance).

DETAILED DESCRIPTION:
The purpose of the Family Help Sleep Program is to deliver, primary care mental health services to children and their families in the comfort and privacy of their own home. Approximately 80 children (6-12 years of age)suffering from mild to moderate sleep onset latency and/or bedtime resistance will be randomized.

The intervention is delivered from a distance, using an educational handbook and telephone consultation with a trained paraprofessional "coach" who is supervised by a licensed health care professional. The telephone coach delivers consistent care based on written protocols, with on-going evaluation by a professional team.

ELIGIBILITY:
Inclusion Criteria:

* children 5-12 years of age
* attending grades primary-6 (Elementary School)
* sleep onset latency and/or bedtime resistance
* speak and write English
* provides parental authorization
* has access to telephone in home

Exclusion Criteria:

* any mental health disease with the exclusion of disruptive behavior disorder
* neurological conditions
* moderate to severe cognitive impairment
* has received a behavioral intervention for sleep difficulties in the past 6 months
* nocturnal enuresis
* sleep apnea
* co-sleeping

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2005-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Child Sleep Habits Questionnaire | baseline, 2months (end of treatment) & 6 month follow-up

SECONDARY OUTCOMES:
Sleep diary | daily during treatment; on follow-up at 2 & 6 MONTHS post randomization
Actigraph recordings | daily during treatment; baseline, 2 & 6 months follow-up
Child Behaviour Checklist (CBCL) | baseline, 2months (end of treatment) & 6 month follow-up
Satisfaction scale (researcher developed) | end of treatment
Parenting Stress Index | baseline, 2months (end of treatment) & 6 month follow-up
Child Health Questionnaire | baseline, 2months (end of treatment) & 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Penny Corkum, PhD., Principal Investigator — IWK Health Centre and Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate summary data would be made available but not individual data.

REFERENCES:
- [Background] Corkum P, Lingley-Pottie P, Davidson F, McGrath P, Chambers CT, Mullane J, Laredo S, Woodford K, Weiss SK. Better Nights/Better Days-Distance Intervention for Insomnia in School-Aged Children With/Without ADHD: A Randomized Controlled Trial. J Pediatr Psychol. 2016 Jul;41(6):701-13. doi: 10.1093/jpepsy/jsw031. Epub 2016 May 16. PMID 27189687